CLINICAL TRIAL: NCT04335656
Title: Reducing Innate Inflammation in New Onset Type 1 Diabetes With Lactiplantibacillus Plantarum
Brief Title: Reducing Innate Inflammation in New Onset Type 1 Diabetes
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Susanne Cabrera, Principal Investigator, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1560525
Record Dates: First submitted 2020-03-27; First posted 2020-04-06 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes; type1diabetes; Type 1 Diabetes Mellitus
Keywords: New onset; Newly diagnosed; Recent onset; Probiotic; Lactiplantibacillus plantarum; Lp299v
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, 2:1 randomly assigned
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Subjects will be randomized to the treatment or placebo group. The treatment is a capsule taken by mouth once a day for 6 months.
  Interventions: Dietary Supplement: Lactiplantibacillus plantarum
- Placebo Group (Placebo Comparator): Subjects will be randomized to the treatment or placebo group. The placebo is a capsule taken by mouth once a day for 6 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactiplantibacillus plantarum — Probiotic capsule in powder form, which can be swallowed or opened and contents sprinkled on cold foods or beverages
  Other Names: Lp299v
  Arms: Treatment Group
Other: Placebo — Placebo capsule in powder form, which can be swallowed or opened and contents sprinkled on cold foods or beverages
  Arms: Placebo Group

SUMMARY:
This study aims to determine whether Lactiplantibacillus plantarum 299v (Lp299v) supplementation will reduce systemic inflammation and prolong residual beta cell function in individuals newly diagnosed with Type 1 diabetes. The investigators hypothesize that probiotic-induced alterations in the intestinal microbiota may favorably alter the post-onset disease state.

DETAILED DESCRIPTION:
For individuals newly diagnosed with Type 1 diabetes, this clinical trial will assess whether probiotic supplementation has efficacy in reducing the endogenous systemic innate inflammatory state known to exist in newly diagnosed Type 1 diabetes and whether this reduction correlates with preservation of endogenous insulin production as measured by stimulated C-peptide during mixed meal tolerance testing (MMTT). The innate inflammatory state will be measured by plasma-induced transcriptional assay and quantified as a composite inflammatory index. Mixed meal tolerance testing is the gold standard measure of endogenous insulin production. During this test, serial blood c-peptide levels are collected over 2 hours in response to challenge with a nutritional drink containing a mix of protein, fat, and carbohydrate and the C-peptide area under the curve is calculated.

Using a randomized, placebo-controlled design, the investigators will measure changes in systemic inflammation (primary outcome) and beta cell function (secondary outcome) after six months of daily treatment with either Lp299v supplementation or placebo. These measures of plasma-induced transcriptional assay and MMTT will be related to markers of beta cell stress, the composition of the gut microbiota, analysis of the plasma metabolome, and levels of microbial antigen exposure.

ELIGIBILITY:
Inclusion Criteria:

1. ≤ 100 days from T1D diagnosis based on ADA criteria
2. > 21 days from T1D diagnosis or metabolically stable per study physician assessment
3. Males and females 3-45 years of age, inclusive, at time of screening visit
4. Peak MMTT stimulated C-peptide ≥ 0.2 nmol/L
5. Positive for at least 1 diabetes autoantibody (excluding mIAA in those who have received ≥ 2 weeks of exogenous insulin therapy) either through clinically obtained labs at time of diagnosis or as obtained at the screening visit
6. Females of child-bearing potential (defined as any female who has reached menarche (first menses), excluding those who have had a hysterectomy or are post-menopausal and must be willing to use effective birth control (which may include abstinence)) from screening visit until final study visit
7. Willing and able to give informed consent or have parent or legal guardian provide informed consent if the subject is < 18 years of age

Exclusion Criteria:

1. Probiotic supplement use within the past month
2. Antibiotic use within the past month
3. Concurrent or recent (within the past 30 days of screening) use of non-insulin therapies aimed to control hyperglycemia
4. Females who are pregnant or lactating
5. Chronic inflammatory or autoimmune disease with exception of stable thyroid disease
6. Uncontrolled celiac disease (i.e., consuming gluten) or actively being evaluated for possible celiac disease (i.e., clinically obtained tissue transglutaminase IgA titers above reference range, being referred to gastroenterology for possible endoscopy, etc.)
7. Use of glucocorticoids or other immunosuppressive agents within 30 days of screening MMTT
8. Use of medications known to influence glucose tolerance
9. Dairy allergy
10. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results.

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in composite inflammatory index after probiotic supplementation | 5 years (duration of study)
  Investigators will examine the effect of probiotic supplementation on the endogenous innate inflammatory state in youth newly diagnosed with T1D, as measured by plasma-induced transcription and analyzed using a composite inflammatory index score. The investigators hypothesize that the subjects receiving the probiotic will have less inflammation (as measured by transcriptional analysis) than the participants in the placebo group.

SECONDARY OUTCOMES:
Rate of stimulated C-peptide Area Under the Curve (AUC) decline after probiotic supplementation | 5 years (duration of study)
  Investigators will examine the rate of C-peptide decline, as measured by C-peptide AUC in youth newly diagnosed with T1D. The investigators hypothesize that the subjects receiving the probiotic for 6 months will have a slower rate of decline than the subjects in the placebo group.
Markers of beta cell function | 5 years (duration of study)
  Investigators will examine the effect of probiotic supplementation on beta cell function by measuring proinsulin levels, ratio of proinsulin to C-peptide and islet amyloid polypeptide to pro-islet amyloid polypeptide ratio.
Microbial composition as measured by 16s rRNA sequencing | 5 years (duration of study)
  Investigators will examine the effect of probiotic supplementation using 16s rRNA sequencing to determine the composition of the intestinal microbiota. Investigators hypothesize the composition of the intestinal microbiota will differ before and after treatment with probiotic supplementation.
Markers of systemic microbial antigen exposure | 5 years (duration of study)
  Gut leakiness will be measured by examining the levels of microbial antigens in the plasma before and after treatment and correlating these antigen levels with the changes in the composition of the gut bacteria. It is hypothesized that changes in antigen levels and gut bacteria will only be seen in the participants receiving the probiotic. It is further hypothesized that those with the greatest reduction in antigens will have the most significant changes in gut bacteria composition.
Regulatory T cell abundance and activity by flow cytometry | 5 years (duration of study)
  Investigators will examine the effect of probiotic supplementation on regulatory T cell abundance and activity.
Monocyte abundance and activity by flow cytometry | 5 years (duration of study)
  Investigators will examine the effect of probiotic supplementation on monocyte abundance and activity.
scRNA-seq analyses of peripheral blood mononuclear cells | 5 years (duration of study)
  Investigators will examine the effect of probiotic supplementation on peripheral blood mononuclear cells using single cell RNA sequencing analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No